CLINICAL TRIAL: NCT06496854
Title: Prescribing Lorazepam for IUD Insertion: Pilot Feasibility Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to coordinate logistics
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0655; A532014 (Other: UW Madison); Protocol Version 6/5/2024 (Other: UW Madison)
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Pain; IUD
Keywords: IUD insertion
MeSH Terms: conditions — Pain | interventions — Lorazepam; Ibuprofen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lorazepam administration prior to IUD insertion procedure (Experimental)
  Interventions: Drug: Lorazepam 1 mg; Drug: Ibuprofen 800 mg

INTERVENTIONS:
Drug: Lorazepam 1 mg — 1 mg oral lorazepam, a sedative used to relieve anxiety
Drug: Ibuprofen 800 mg — 800 mg ibuprofen, Nonsteroidal anti-inflammatory drug to treat pain

SUMMARY:
The objective of this pilot study is to discuss the feasibility of prescribing lorazepam prior to IUD insertion and of measuring effect of lorazepam on anxiety and pain with Intrauterine Device (IUD) insertion. The target population for this study will be 25 adult participants scheduled for an IUD insertion at a UW Family Medicine residency clinic. Participants will be followed for 1 appointment visit.

DETAILED DESCRIPTION:
The purpose of the research is to evaluate the feasibility of prescribing lorazepam and measuring its effect on anxiety and pain with IUD insertion. The descriptive data from this study will be used to offer guidance for how to implement a larger scale study in the future.

Primary endpoint: Assess preliminary differences in pain and anxiety scores pre-IUD insertion and post-IUD insertion using a Mann-Whitney U test. Participants will score their anxiety and pain levels pre-procedure and post-procedure using a 10cm visual analogue scale. This will be a one arm trial where all subjects will receive 1mg lorazepam and 800mg ibuprofen prior to the procedure.

Secondary endpoints

* Discuss if there was a difference in pain and anxiety scores among nulliparous (no previous childbirths) and multiparous (one or more previous childbirths) participants.
* Summarize recruitment rates, adherence to lorazepam prescription, completion rates of questionnaires and scales
* Discuss participant's experiences with taking lorazepam and participating in the study
* Assess investigator's experience with the trial via a focus group

ELIGIBILITY:
Inclusion Criteria:

* Participants who undergo IUD insertion and complete the visual analogue scales to rate their anxiety and pain level prior to the procedure and after the procedure.
* Participants must have a driver take them to their appointment if they take lorazepam prior to their arrival at the clinic.
* Participants must have a driver take them home after the procedure as well.
* Participants must consent to email communication since they will sign the consent forms electronically

Exclusion Criteria:

* Participants who do not show up for their appointment.
* Participants who receive cervical blocks or other analgesic method during IUD insertion.
* Participants who have a history of substance use disorder.
* Participants who are taking medications with a central nervous system (CNS) depressant effect (ex: opioids, benzodiazepines).
* Participants who are not able to sign an electronic consent form.
* Participants who do not have a driver to take them to their appointment and to take them home after the procedure.
* Participants who do not agree to sign consent forms electronically.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale for Pain | before and after the procedure (up to 1 hour)
  Participant will be asked to rate their pain on a scale of 0 (no pain) to 10 (severe pain).
Visual Analogue Scale for Anxiety | before and after the procedure (up to 1 hour)
  Participant will be asked to rate their anxiety on a scale of 0 (no anxiety) to 10 (severe anxiety).

SECONDARY OUTCOMES:
Mean Pain Scores for Nulliparous and Multiparous Participants | before and after the procedure (up to 1 hour)
  Comparison of mean pain scores between participants that have never had childbirth to those who have.
Mean Anxiety Scores for Nulliparous and Multiparous Participants | before and after the procedure (up to 1 hour)
  Comparison of mean anxiety scores between participants that have never had childbirth to those who have.
Number of Participants Recruited | up to 2 months (estimated time period of recruitment)
  Feasibility will in part be measured with recruitment rates.
Number of Participants with lorazepam prescription adherence | up to 2 months (estimated time period of recruitment)
  Feasibility will in part be measured with adherence rates.
Number of Participants Who Completed All Surveys | up to 2 months (estimated time period of recruitment)
  Feasibility will in part be measured with survey completion rates.
Qualitative Measure: Participant Experience | post-procedure (up to 1 hour)
  Participants will be asked questions about their experience taking lorazepam and to provide feedback about the study. Participant answers will be coded and themed to report as participant counts.

CONTACTS AND LOCATIONS:
Overall Officials: Jensena Carlson, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW Family Medicine Residency Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No